CLINICAL TRIAL: NCT06030102
Title: Voiding Log and Fluid Intake Habits Among Young Healthy Population
Brief Title: Voiding Log and Fluid Intake Habits
Status: Completed | Type: Observational
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 25
Record Dates: First submitted 2020-11-18; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2020-11

CONDITIONS: Young Healthy Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy young population

SUMMARY:
Health practitioners usually instruct patients with complaints of urinary incontinence and urinary tract infection regarding voiding and fluid intake habits. However poor drinking habits develop early in life, even prior to the symptoms presentation. Little is known about the voiding habits and fluid intake routine among healthy young population. The current study aims to assess the habits of drinking and voiding log among such population.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female Adolescent healthy population

Exclusion Criteria:

* History of incontinence Symptoms of urinary tract infection History of any pelvic floor disorder

Ages: 24 Years to 38 Years | Sex: All
Age Groups: Adult
Study Population: Population comprises of both male and females. Young Healthy population aged between 24 to 38 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Fluid intake | 1 month
  amount of cups taken per day
Voiding | 1 month
  voiding diary

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr.Javed Akram, MBBS,FRCP,MRCP, Study Chair — University of Health Sciences Lahore Pakistan; Dr. Irum Shah, Study Director — Penn Medicine Healthcare New Jersey, USA; Dr. Muhammad Sheraz Alam, Principal Investigator — Lahore College of Physical Therapy, LM&DC Lahore Pakistan; Dr. Maleeha Fuad, Principal Investigator — Lahore College of Physical Therapy, LM&DC Lahore Pakistan
Locations (1):
- University of Health Sciences, Lahore, Punjab Province, Pakistan